CLINICAL TRIAL: NCT06253481
Title: Cardiovascular Diseases: Investigating the Risk Factors and Clinical Features Using Multi-omics Technologies
Brief Title: Genetics of Cardiovascular Disease
Acronym: GCVD
Status: Recruiting | Type: Observational
Sponsor: Center for Strategic Planning, of the Federal Medical and Biological Agency (Other)
Collaborators: National Medical Research Center for Cardiology, Ministry of Health of Russian Federation (Other Government)
Responsible Party: Sponsor
Other Study IDs: Cardiogen
Record Dates: First submitted 2024-02-02; First posted 2024-02-12 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Atherosclerosis; Coronary Heart Disease; Myocardial Infarction; Atrial Fibrillation
Keywords: Atherosclerosis; coronary heart disease; myocardial infarction; atrial fibrillation; polygenic risk panel; multi-omics study
MeSH Terms: conditions — Atherosclerosis; Coronary Disease; Myocardial Infarction; Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole blood, serum
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group I: patients diagnosed with various types of ASCVD: Group I: Patients diagnosed with various types of ASCVD (> 50% stenosis caused by atherosclerotic plaque) of various vascular beds (coronary vessels, carotid arteries, mesenteric arteries, lower extremities, and kidneys) (case; n=6500).
- Group II: patients with no clinically significant ASCVD (control, n=3500): Group II: patients with no ultrasound/ angiography findings of ASCVD (control, n=3500)

SUMMARY:
Participants are being recruited at the inpatient department of the National Medical Research Center of Cardiology on a 'all-comers' basis. The enrolled participants will be divided into the main group (diagnosed with atherosclerotic cardiovascular disease (ASCVD)) and control (not diagnosed with ASCVD). The participants will have whole blood and serum collected at enrollment for further biobanking. A genome-wide association study will be carried out to determine the genetic determinants associated with atherosclerosis, coronary heart disease, acute coronary syndrome, etc., including a search for pathogenic variants.

DETAILED DESCRIPTION:
This is a non-interventional case-control study aimed at identifying the genetic markers associated with various ASCVD types or with the protective effect against them. Participants are being recruited at the National Medical Research Center for Cardiology of the Ministry of Health of Russia. The study will comprise at least 10,000 participants, 1 non-ASCVD patient per 2 ASCVD patients. The recruitment period started in September 2021 and will continue till December 2023. The study will be conducted for 29 months. Observation will be carried out throughout the study.

The participants of this study will be selected from the patients of the inpatient treatment at the National Medical Research Center of Cardiology. This study procedures will have no effect on the diagnostic and therapeutic procedures implemented by the attending physicians, based on the protocols and recommendations adopted in the Russian Federation.

All participants will be divided into 2 groups:

1. Patients with severe atherosclerosis (≥ 50% stenosis caused by atherosclerotic plaque) of various vascular beds (coronary vessels, carotid arteries, mesenteric arteries, lower extremities, and kidneys)
2. Control group without clinically significant atherosclerotic lesions (≤49% stenosis).

In each group, the known risk factors and the genetic determinants of ASCVD will be investigated. Based on the results of the analysis of all factors under consideration, the study should yield a panel of ASCVD markers.

ELIGIBILITY:
Inclusion criteria:

1. At least 18 years of age;
2. Informed consent;
3. An in-patient available for a comprehensive assessment for ASCVD.

Exclusion criteria:

1. Refusal to participate;
2. Positive/negative ASCVD impossible to confirm;
3. HIV, syphilis, hepatitis B and C;
4. Any other criteria deemed reasons for exclusion by the Principal Investigator

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: In-patients of the National Medical Research Center for Cardiology from various regions of the Russian Federation.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2021-11-24 (Actual); Primary Completion 2025-11-24 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Identification of the genetic determinant associated with ASCVD, coronary heart disease, and myocardial infarction; 1) Identification of the genetic determinant associated with ASCVD, coronary heart disease, and myocardial infarction | up to 24 month
Determining the frequency of the pathogenic variants in the study cohort, including in the participants with the early onset of atrial fibrillation, myocardial infarction, and carotid artery disease, etc. | up to 24 month

CONTACTS AND LOCATIONS:
Overall Officials: Marat V. Ezhov, M.D., Ph.D, Principal Investigator — National Medical Research Center of Cardiology named after Academician E.I. Chazov, Ministry of Health of the Russian Federation
Locations (2):
- Russia (2):
  - National Medical Research Center of Cardiology named after Academician E.I. Chazov, Ministry of Health of the Russian Federation, Moscow
  - Federal State Budgetary Institution Centre for Strategic Planning and Management of Biomedical Health Risks of the Federal Medical Biological Agency, Moscow

IPD SHARING:
Plan to Share IPD: No